CLINICAL TRIAL: NCT04123197
Title: Mental Stress and Myocardial Ischemia After MI: Sex Differences, Mechanisms and Prognosis
Acronym: MIMS3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Viola Vaccarino, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00113346; 2R01HL109413-05A1 (NIH)
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction
Keywords: Cardiovascular disease; Daily life stressors; Mental stress-induced myocardial ischemia (MSI)
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young Participants with Prior MI (Other): Participants aged 60 or less who experienced a MI within the last 8 months will undergo a stress challenge to assess MSI and will then be followed for 3 years.
  Interventions: Other: Stress Challenge

INTERVENTIONS:
Other: Stress Challenge — The stress challenge will assess how different parts of the body react to stress. Participants will be given no specific details about the contents of the test before administration.

SUMMARY:
The purpose of this study is to look at the link between emotional stress and heart disease in men and women. Taking part in this study involves one clinic visit, one week of at home monitoring, and follow up phone calls every 6 months for 3 years.

DETAILED DESCRIPTION:
In the U.S. and globally, coronary heart disease (CHD) is the number one killer of women. Despite scientific advances, it is unclear whether the pathophysiology of CHD differs between women and men. The study of CHD in women has historically been centered on older women, however, women with early onset CHD are informative for the study of early risk factors and pathophysiology. Furthermore, young women with a myocardial infarction (MI) have emerged as a group in need of special study as this group has higher mortality compared with men of similar age despite less severe disease. These disparities remain unexplained and suggest sex differences in the pathophysiology, risk factors and prognostic factors of acute MI.

The psychosocial sphere is a largely neglected area for CHD prevention in women. Social and emotional exposures mostly beginning early in life (depression, early life adversities, poverty and posttraumatic stress symptoms) are more common in younger women with MI compared with men and community controls. In addition to being more prevalent, it is possible that emotional stress is a stronger risk factor in young women than other groups. A significant challenge, however, is to measure stress in a valid way.

Building on previous work, the current project will clarify sex differences in pathways of risk linking emotional stress to mental stress-induced myocardial ischemia (MSI) and cardiovascular outcomes in young post-MI patients. Within 8 months of MI, 310 patients ≤60 years of age (at the time of the MI), 50% women, will be tested in the lab with a stress challenge to asses MSI using an established protocol with myocardial perfusion imaging. Participants will be monitored at home for 1 week, and then followed for clinical events for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* History of documented MI within the past 8 months
* Age ≤60 at the time of MI

Exclusion Criteria:

* History of unstable angina, MI, or decompensated heart failure in the past month
* Patients deemed to be unsafe to hold anti-ischemic medications before testing (it is standard protocol to hold these meds before imaging studies)
* Systolic blood pressure (SBP) >180 mm Hg or diastolic blood pressure (DBP) >110 mm Hg on the day of the test
* Alcohol or substance abuse (past year), or severe psychiatric disorder other than major depression
* Other serious medical disorders that may interfere with the study results
* Postmenopausal hormone therapy (past 3 months)
* Current psychotropic medications (past month) except anti-depressants
* Pregnancy or breastfeeding (all women will receive a pregnancy test)
* Severe aortic stenosis
* Weight ≥ 360 pounds and/or body mass index (BMI) of 40 or greater (weight limit of the SPECT imaging table)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 311 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Events | 3 Years
  The main outcome will be a composite endpoint of recurrent MI, unstable angina, hospitalization for decompensated heart failure, and cardiovascular (CV) death. A mental stress-induced myocardial ischemia (MSI) status of positive or negative will be the main predictor in regression models.

SECONDARY OUTCOMES:
Myocardial Infarction or Cardiovascular Death | 3 Years
  The number of participants experiencing myocardial infarction or CV death in relation to MSI status (positive or negative).
Cardiovascular Death | 3 Years
  The number of participants experiencing CV death in relation to MSI status (positive or negative).
Total Mortality | 3 Years
  The number of participants experiencing all-cause death in relation to MSI status (positive or negative).
Cardiovascular Events Excluding Heart Failure | 3 Years
  This is a composite endpoint of recurrent MI, unstable angina, or CV death where the number of participants experiencing this endpoint in relation to MSI status (positive or negative) will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Viola Vaccarino, MD, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah AJ, Weeks V, Lampert R, Bremner JD, Kutner M, Raggi P, Sun YV, Lewis TT, Levantsevych O, Kim YJ, Hammadah M, Alkhoder A, Wittbrodt M, Pearce BD, Ward L, Sheps D, Quyyumi AA, Vaccarino V. Early Life Trauma Is Associated With Increased Microvolt T-Wave Alternans During Mental Stress Challenge: A Substudy of Mental Stress Ischemia: Prognosis and Genetic Influences. J Am Heart Assoc. 2022 Mar;11(5):e021582. doi: 10.1161/JAHA.121.021582. Epub 2022 Feb 15. PMID 35167312

DOCUMENTS (1):
  • Informed Consent Form (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT04123197/ICF_000.pdf